CLINICAL TRIAL: NCT00218634
Title: CBT for Depression & Adherence in HIV Methadone Patients
Brief Title: Skills Based Counseling for Adherence and Depression in HIV+ Methadone Patients - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-18603-1; R01DA018603 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Adherence; Depression; Heroin Dependence; Methadone; Motivational Interviewing; Substance-Related Disorders
MeSH Terms: conditions — Depression; Heroin Dependence; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-AD (Experimental): Cognitive behavioral therapy for adherence and depression
  Interventions: Behavioral: CBT-AD
- ETAU (Active Comparator): Enhanced treatment as usual
  Interventions: Behavioral: ETAU

INTERVENTIONS:
Behavioral: CBT-AD — Cognitive behavioral therapy for adherence and depression consisting of 1 session focusing on adherence and 8 sessions consisting of cognitive behavioral therapy for medication adherence and depression.
  Arms: CBT-AD
Behavioral: ETAU — Enhanced treatment as usual consisting of 1 session focused on adherence (the same session as the CBT-AD intervention) and 8 sessions for participants to complete self-reports and collect adherence data.
  Arms: ETAU

SUMMARY:
Patients with HIV, depression, and opioid-dependence are at high risk for poor health outcomes. This is a two-arm randomized controlled trial of cognitive-behavioral therapy for depression and HIV medication adherence in patients with opioid dependence who are receiving methadone maintenance treatment. The project is based on our pilot work with close attention to NIDA guidelines for a staged approach to treatment development and testing (Rounsaville et al., 2001).

Depression is highly comorbid with both HIV infection and with opioid dependence. Depression and substance abuse are both associated with poor adherence to antiretroviral medications. Patients with HIV, depression, and opioid dependence are at high risk for poor health outcomes. Cognitive-behavioral therapy is the most widely studied and efficacious psychosocial intervention for depression; and research by the PI and others has shown that cognitive-behavioral interventions have been successful in promoting adherence to HIV medications.

DETAILED DESCRIPTION:
Symptoms of depression (i.e. low motivation, poor concentration, loss of interest, sad mood, suicidal ideation) that occur in the context of substance abuse or dependence can interfere with self-care behaviors necessary for maintaining HIV care, as well as interfere with potential benefit from an intervention that focuses on adherence alone. We hypothesize that teaching skills to cope with depression will improve the outcome from an adherence intervention to promote healthier living with HIV, in HIV+ opioid dependent individuals in methadone maintenance treatment.

Overview of Research Plan. Patients who are HIV positive and who are receiving methadone maintenance for opioid dependence will be randomized to treatment with either: (1) CBT, a combination of CBT for depression and HIV medication adherence, including a single session intervention for HIV medication adherence (Life-Steps, Safren et al., 2001) in conjunction with physician feedback regarding baseline study assessments or (2) the single session intervention for HIV medication adherence (Life-Steps, Safren et al., 2001) in conjunction with physician feedback regarding baseline study assessments. Participants will be followed for one-year post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* Currently enrolled in methadone maintenance treatment for at least one month
* Current major or subsyndromal depression (subsyndromal depression is defined by major depression that does not meet full diagnostic criteria but with a clinical global impression of severity (CGI-S) of 2 (mildly ill))
* Is prescribed antiretroviral therapy for HIV and therefore under the care of a primary care provider.
* Between the ages of 18 and 65.

Exclusion Criteria:

* Active untreated, unstable, major mental illness (i.e., untreated psychosis or mania), or other Axis I psychiatric disorders (other than depression) that would interfere with the ability to participate (i.e. CGI-S >6)
* Unable or unwilling to provide informed consent.
* Currently in cognitive behavioral therapy for depression.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2005-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Safren, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Safren SA, O'Cleirigh CM, Bullis JR, Otto MW, Stein MD, Pollack MH. Cognitive behavioral therapy for adherence and depression (CBT-AD) in HIV-infected injection drug users: a randomized controlled trial. J Consult Clin Psychol. 2012 Jun;80(3):404-15. doi: 10.1037/a0028208. Epub 2012 Apr 30. PMID 22545737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participants from methadone clinics, remainder from MGH or RIH clinics.
Pre-assignment Details: Participants had to screen for study inclusion/exclusion criteria before randomization.
Period: Overall Study
Arm/Group | CBT-AD | ETAU
Started | 44 | 45
Completed | 36 | 30
Not Completed | 8 | 15
Not completed — Lost to Follow-up | 8 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT-AD | ETAU | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 45 | 89
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.05 (7.34) | 46.67 (7.05) | 46.85 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 27 | 27 | 54
Region of Enrollment [Number; unit: participants]
  United States | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Percent Medication Adherence at 3-month Follow-up Assessment
Description: Post-treatment assessment in adherence to HIV medication. Doses taken were assessed by downloading information from the electronic pill cap and corroborated by participant self-report. Adherence was calculated as the number of doses taken over the time period divided by the number of doses prescribed.
Time Frame: 3-month assessment
Population: We used hierarchical linear modeling (HLM) methods and intent to treat for all randomized participants.
Measure: Mean (Standard Deviation); unit: percent (doses taken/doses prescribed)
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
percent (doses taken/doses prescribed) | 79.02 (23.23) | 73.66 (25.15)
Statistical Analysis 1: Comparison: CBT-AD vs ETAU; We used HLM with weekly visit data for the acute outcome. There were, therefore, 11 time points used; Test type: Superiority or Other; p < .05, HLM

2. Secondary Outcome: Clinician-assessed Depression Rating at 3 Month Follow-up Assessment
Description: Depression was assessed using the Montgomery-Asberg Depression Rating Scale (MADRS) by a clinical interviewer blind to participants' study condition. The scale ranges from 0 to 60 with 7-19 indicating mild depression and 20-34 indicating moderate depression.
Time Frame: 3 month follow-up
Population: We used intent to treat for all data analysis.
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Cognitive Behavioral Therapy for Adherence and Depression: Cognitive behavioral therapy focusing on treating depression and adherence to medication (CBT-AD).
- Enhanced Treatment as Usual: Enhanced treatment as usual (ETAU).
Arm/Group | Cognitive Behavioral Therapy for Adherence and Depression | Enhanced Treatment as Usual
Number analyzed (Participants) | 44 | 45
Units on scale | 17.02 (10.62) | 22.7 (10.19)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy for Adherence and Depression vs Enhanced Treatment as Usual; Test type: Superiority or Other; p < .05, GLM and HLM — GLM - CBT-AD would be superior to ETAU at post. HLM - CBT-AD would be superior to CBT-AD at follow ups

3. Secondary Outcome: HIV Viral Load at 12-month Follow-up Assessment
Description: HIV plasma RNA (log HIV viral load)at the 12-month follow-up assessment.
Time Frame: 12-month follow-up assessment
Population: We used intent to treat for all data analysis.
Measure: Log Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
log10 copies/mL | 2.203 (0.687) | 2.177 (0.820)

4. Secondary Outcome: CD4+ Lymphocyte Count at 12-month Follow-up Assessment.
Description: CD4+ lymphocyte cell count at 12-month follow-up assessment.
Time Frame: 12-month follow-up assessment
Population: We used intent to treat for all data analysis.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
cells/mm^3 | 452.94 (235.00) | 502.33 (314.19)
Statistical Analysis 1: Comparison: CBT-AD vs ETAU; follow up analysis revealed that CD4, over time, significantly improved over control when covarying out baseline levels; Test type: Superiority or Other; p < .05, HLM — CD4 would be more improved in the treatment condition

5. Primary Outcome: Percent Medication Adherence at 12-month Follow-up Assessment
Description: Follow-up assessment in adherence to HIV medication. Doses taken were assessed by downloading information from the electronic pill cap and corroborated by participant self-report. Adherence was calculated as the number of doses taken over the time period divided by the number of doses prescribed.
Time Frame: 12-month follow-up assessment
Population: We used intent to treat for all data analysis.
Measure: Mean (Standard Deviation); unit: percent (doses taken/doses prescribed)
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
percent (doses taken/doses prescribed) | 64.49 (31.34) | 61.11 (34.94)

6. Secondary Outcome: Clinician-assessed Depression at 12-month Follow-up Assessment
Description: as for outcome 2
Time Frame: 12-month follow-up assessment
Population: We used intent to treat for all data analysis.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
Units on scale | 15.28 (9.22) | 20.00 (10.97)

7. Secondary Outcome: HIV Viral Load at 3-month Follow-up Assessment
Description: HIV plasma RNA (log HIV viral load)at the 3-month follow-up assessment.
Time Frame: 3-month assessment
Population: We used intent to treat for all data analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/mL"
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
log10 copies/mL" | 2.349 (0.928) | 2.044 (0.509)

8. Secondary Outcome: CD4+ Lymphocyte Count at 3-month Follow-up Assessment.
Description: CD4+ lymphocyte cell count at 3-month follow-up assessment.
Time Frame: 3-month assessment
Population: We used intent to treat for all analysis.
Measure: Mean (Standard Deviation); unit: cells/mm3
Arm/Group | CBT-AD | ETAU
Number analyzed (Participants) | 44 | 45
cells/mm3 | 380.97 (266.62) | 539.29 (293.61)

ADVERSE EVENTS:
Time Frame: Adverse events are reported for a given participant for the time that participant was enrolled in the trial (roughly 1 year).
Description: Serious adverse events reported include those that were study related.
Arm/Group | CBT-AD | ETAU
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 0/44 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No